CLINICAL TRIAL: NCT01982864
Title: Pharmacokinetics of an Aminoglycoside in Hemodialysis Patients.
Acronym: DIAMS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: I12008 DIAMS
Record Dates: First submitted 2013-10-31; First posted 2013-11-13 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis
Keywords: Aminoglycosides; hemodialysis; clinical pharmacokinetics; pharmacokinetic modelling; Bayesian estimation; Necessity; of the treatment; gentamicin
MeSH Terms: interventions — Gentamicins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hemodialysis patients (Experimental): The administration of gentamicin at the beginning of the hemodialysis.
  Interventions: Drug: Gentamicin

INTERVENTIONS:
Drug: Gentamicin — The decision to introduce the antibiotic is made during a session or between two sessions according to both the clinicians usual procedure.
  Depending on the number of injections, 8 to 10 blood samples will be drawn per patient. Clinical and biological data will be concomitantly collected (e.g., hemodialysis session duration, creatinine clearance…).
  The number of blood sampling and the time schedule will be adapted to the prescription and the possible follow-up of the treatment after the first injection. Whatever the time is between the first injection and the following dialysis session, a sampling will be performed 30 minutes after the end of the injection (T1), 8h after the end of the injection (T2), juste before (TAD), in the middle (TMD) and at the end of the dialysis (TFD).

SUMMARY:
Aminoglycosides are widely used for the treatment of Gram-negative bacilli and Staphylococcus aureus infections because of their effectiveness and low cost. Nevertheless, many aspects of their optimal use in hemodialysis patients remain unsolved and little is known about their pharmacokinetics in this context. The current practice for prescribing aminoglycosides to these particular patients consists in giving after each hemodialysis session about half the dose usually given to patients with normal renal function.

However, theoretical considerations and emerging clinical data suggest that this may not be the most beneficial dosing regimen as efficient peak concentrations are often not attained and the occurrence of ototoxicity and nephrotoxicity is still frequent.

DETAILED DESCRIPTION:
Recent evidence about the pharmacokinetics and pharmacodynamics of aminoglycosides strongly supports administration of aminoglycosides before, rather than after, hemodialysis. Therapeutic drug monitoring using pharmacokinetic modeling is currently used in non-hemodialysis patients. However, the PK tools employed are not suitable to dialysis patients.

For aminoglycosides, the ratio of peak to Minimal Inhibitory Concentration (MIC) has been shown to be the parameter that best correlates with clinical efficacy, whilst prolonged exposure to high concentrations have been related to either nephrotoxicity or ototoxicity. Additionally, aminoglycosides are mostly excreted as unchanged drugs in urine and their clearance is directly proportional to the glomerular filtration rate. The elimination half-life of aminoglycosides is approximately 1.5-3 hours in adults with normal renal function, but is greatly prolonged up to 36-70 hours in patients with end-stage renal failure. In a standard patient, aminoglycosides are administered as a single dose, over a short time interval, to obtain an elevated blood peak concentration (the effective level). The next injection is not administered before 24 hours, to allow the patient to wash out the aminoside and to minimize the residual blood concentration (the toxic level). The aim here is to maximize the peak concentration during a fair amount of time (by repeating the peaks) and to minimize the overall drug exposure, responsible for the toxicity.

For the renal impaired patient, our hypothesis is that the hemodialyzer can be regarded as a kidney. Thus, the administration of the aminoside at the beginning of the hemodialysis could lead to profiles of elimination comparable to those observed in normorenal patients.

The research aims at performing a population pharmacokinetic (POPPK) study of gentamicin when given to hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* age upper to 18 years
* Patients hospitalized in the "Service de Néphrologie - Hémodialyse, Transplantations, CHU de Limoges"
* Patients requiring chronic hemodialysis
* Patients requiring a treatment by aminoglycosides
* Patients willing to give their written informed consent for their participation to the study
* Patients affiliated to the French social security system or equivalent

Exclusion Criteria:

* Patients under legal protection
* Patients unable or unwilling to provide informed consent and not under legal protection
* Patients deprived of liberty
* Contraindications to gentamicin
* Pregnant or breast-feeding women or women of childbearing potential without efficient contraception (based on declaration)
* Patients with any altered mental status or any psychiatric condition that would interfere with the understanding of the study
* Patients enrolled in another clinical trial testing drugs or therapeutic strategies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Concentration curves of gentamicin | 1 week
  The research aims at performing a population pharmacokinetic (POPPK) study of gentamicin when given to hemodialysis patients.
  The ability to describe the concentration curves versus time (Biais (%) between the observed concentrations and the concentrations predicted by the model).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre MARQUET, MD, Principal Investigator — CHU LIMOGES
Locations (2):
- France (2):
  - CHU LIMOGES - Laboratoire de Pharmacologie, Limoges
  - CHU LIMOGES - Service Néphrologie, Limoges

REFERENCES:
- [Result] Franck B, Monchaud C, Saint-Marcoux F, Rerolle JP, Allard J, Allot V, Marquet P, Essig M, Woillard JB. Population pharmacokinetics of gentamicin in haemodialysis patients: modelling, simulations and recommendations. Eur J Clin Pharmacol. 2020 Jul;76(7):947-955. doi: 10.1007/s00228-020-02867-3. Epub 2020 May 1. PMID 32358683